CLINICAL TRIAL: NCT02285868
Title: ATI Evidence-based Guide Investigating Clinical Services: Rehabilitation and Physical Therapy Patient Outcomes Registry
Brief Title: ATI Evidence-based Guide Investigating Clinical Services
Acronym: AEGIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ATI Holdings, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ATI EGIS01012015
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Spine Osteoarthritis; Shoulder Impingement Syndrome; Knee Osteoarthritis; Hip Osteoarthritis; Osteoarthritis; Carpal Tunnel Syndrome; Fracture; Sprain
Keywords: Orthopedic rehabilitation; Rehabilitation outcomes; Physical therapy; Physical therapy outcomes
MeSH Terms: conditions — Osteoarthritis, Spine; Shoulder Impingement Syndrome; Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis; Carpal Tunnel Syndrome; Fractures, Bone; Sprains and Strains

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Arm, Shoulder and Hand injuries: Pre- and post-treatment outcomes of care as measured by the DASH (Disabilities of the Arm, Shoulder and Hand) via physical therapy
- Lumbar spine injuries: Pre- and post-treatment outcomes of care as measured by the Modified Oswestry (lumbar spine) via physical therapy
- Knee injuries: Pre- and post-treatment outcomes of care as measured by the Knee Outcome Survey via physical therapy
- Foot and ankle injuries: Pre- and post-treatment outcomes of care as measured by the Foot & Ankle Ability Measure via physical therapy
- Hip and lower extremity injuries: Pre- and post-treatment outcomes of care as measured by the Lower Extremity Functional Scale via physical therapy
- Neck injuries: Pre- and post-treatment outcomes of care as measured by the Neck Disability Index Questionnaire via physical therapy

SUMMARY:
The investigators goal is to provide a mechanism that allows for a better understanding of patient outcomes following rehabilitation. This includes functional outcomes measured by standardized and validated tools from the published literature. It incorporates comorbidities and patient demographic characteristics. It includes measures of general health as well along with activities of daily living and behavioral health aspects. Measures of quality and satisfaction and use of Net Promoter Scores also are included. All of these components come together to form a remarkably comprehensive picture of patients and their associated outcomes. This is a unique milestone in rehabilitative care and will act to inform and direct evidence-based approaches and treatment guidelines.

Data are collected via the investigators proprietary electronic medical record system and are synthetic to the clinical process-that is, the data are collected in real-time with patients and the scores are immediately provided to the treating therapist as well as archived for later Registry and scientific use. Subsequent reporting can be risk adjusted to any variable collected which yields robust insights as to idiopathic patient conditions. However, no PHI information will be available.

DETAILED DESCRIPTION:
This is a retrospective, longitudinal, observational registry study to provide a unique and effective mechanism to acquire real-world data on patients receiving physical therapy in a variety of settings, regardless of disorder being treated.

In addition to the standard visit/data collection, patients in the AEGIS™ Registry will also be asked to complete a Quality of Life Questionnaire (SF-12) and a standardized functional outcome instrument. Generally, the following will be available:

Patient Initial Assessment for Physical Therapy:

* De-identified Protected Health Information in accordance to 45 CFR 164.514
* Diagnosis and history Baseline functional outcome measure(s)
* DASH (Disabilities of the Arm, Shoulder and Hand)
* Modified Oswestry (lumbar spine)
* Knee Outcome Survey
* Foot & Ankle Ability Measure
* Lower Extremity Functional Scale
* Neck Disability Index Questionnaire
* Pain rating
* Global Rating of Change Scale
* Baseline Quality of Life Questionnaire (SF-12)

Patient Start of Care:

* Patient information (age, BMI, sex, de-identified Protected Health Information in accordance to 45 CFR 164.514)
* Medical/surgical history
* Therapy review (diagnosis, therapy)
* Treatment plan

Ongoing Patient Assessment:

* De-identified Protected Health Information in accordance to 45 CFR 164.514
* Treatment plan update(s)
* Concurrent (every 10th visit) administration of functional outcome measure(s)
* Concurrent (every 10th visit) administration of Quality of Life Questionnaire (SF-12)
* Patient Satisfaction
* Mailed to discharged patient within a week of discharge from physical therapy with a self-addressed, stamped return envelope Insurance Information
* Insurance carriers
* Insurance coverage

ELIGIBILITY:
Inclusion Criteria:

* Anyone (over the age of 16, all sexes, and diagnoses) receiving physical therapy

Exclusion Criteria:

* Is under age 16
* Has no more than 2 visits/treatment experiences
* Is seen only for an evaluation

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting ith orthopedic rehabilitation needs
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2014-11; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional status | 60 days

SECONDARY OUTCOMES:
Change in global health status | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stout, PsyD, Principal Investigator — ATI and College of Medicine, University of Illinois at Chicago
Locations (1):
- ATI, Bolingbrook, Illinois, United States

REFERENCES:
- [Background] Institute of Medicine, Committee on Quality of Health Care in America. Crossing the Quality Chasm: A new Health System for the 21st Century. Washington, DC: National Academy; 2001.
- [Background] Straus SE, Glasziou P, Richardson WS, Haynes RB. Evidence-Based Medicine: How to Practice and Teach EBM. 4th ed. Edinburgh: Elsevier Churchill Livingstone; 2011.
- [Background] Evidence-Based Medicine Working Group. Evidence-based medicine. A new approach to teaching the practice of medicine. JAMA. 1992 Nov 4;268(17):2420-5. doi: 10.1001/jama.1992.03490170092032. No abstract available. PMID 1404801
- [Background] Bithell C. Evidence-based physiotherapy: Some thoughts on "best evidence". Physiotherapy. 2000; 86: 58-60.
- [Background] Stillwell SB, Fineout-Overholt E, Melnyk BM, Williamson KM. Evidence-based practice, step by step: asking the clinical question: a key step in evidence-based practice. Am J Nurs. 2010 Mar;110(3):58-61. doi: 10.1097/01.NAJ.0000368959.11129.79. PMID 20179464
- [Background] Bernhardsson S, Larsson ME. Measuring evidence-based practice in physical therapy: translation, adaptation, further development, validation, and reliability test of a questionnaire. Phys Ther. 2013 Jun;93(6):819-32. doi: 10.2522/ptj.20120270. Epub 2013 Feb 21. PMID 23431214
- [Background] Wilt TJ. Uncertainty in prostate cancer care: the physician's role in clearing the confusion. JAMA. 2000 Jun 28;283(24):3258-60. doi: 10.1001/jama.283.24.3258. No abstract available. PMID 10866876
- [Background] Woolf SH. The need for perspective in evidence-based medicine. JAMA. 1999 Dec 22-29;282(24):2358-65. doi: 10.1001/jama.282.24.2358. PMID 10612327
- [Background] Croft P, Malmivaara A, van Tulder M. The pros and cons of evidence-based medicine. Spine (Phila Pa 1976). 2011 Aug 1;36(17):E1121-5. doi: 10.1097/BRS.0b013e318223ae4c. No abstract available. PMID 21629165
- [Background] Sterne JA, Davey Smith G. Sifting the evidence-what's wrong with significance tests? BMJ. 2001 Jan 27;322(7280):226-31. doi: 10.1136/bmj.322.7280.226. No abstract available. PMID 11159626
- [Background] Risch NJ. Searching for genetic determinants in the new millennium. Nature. 2000 Jun 15;405(6788):847-56. doi: 10.1038/35015718. PMID 10866211
- [Background] Jasny BR, Chin G, Chong L, Vignieri S. Data replication & reproducibility. Again, and again, and again .... Introduction. Science. 2011 Dec 2;334(6060):1225. doi: 10.1126/science.334.6060.1225. No abstract available. PMID 22144612
- [Background] Seligman MEP, Levant R. Managed care policies rely on inadequate science. Prof Psychol Res Pr. 1998; 29: 211-212.
- [Derived] Lutz AD, Brooks JM, Chapman CG, Shanley E, Stout CE, Thigpen CA. Risk Adjustment of the Modified Low Back Pain Disability Questionnaire and Neck Disability Index to Benchmark Physical Therapist Performance: Analysis From an Outcomes Registry. Phys Ther. 2020 Apr 17;100(4):609-620. doi: 10.1093/ptj/pzaa019. PMID 32285130